CLINICAL TRIAL: NCT00482118
Title: A Hospital-Based Case-Control Study of Non-Smoking Women in Xuan Wei and Fu Yua, China: PAH Exposure, Genetic Susceptibility, and Lung Cancer
Brief Title: Smoky Coal Exposure, Genetic Susceptibility, and Lung Cancer in Non-Smoking Women in China
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999906092; 06-C-N092; NCT00341926 (obsolete NCT alias)
Record Dates: First submitted 2007-06-01; First posted 2007-06-04 (Estimated); Last update posted 2020-11-27 (Actual); Status verified 2020-11

CONDITIONS: Lung Neoplasms
Keywords: Air Pollution; Tumor Markers; Genetic Polymorphisms; Molecular Epidemiology; Environmental Epidemiology
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- Cases: Non smoking women with lung cancer
- Controls: Non smoking women without lung cancer

SUMMARY:
Background:

* Women in Xuan Wei County, China, are almost all non-smokers, yet they have the highest lung cancer rate in that country.
* Non-smoking women in Xuan Wei who use smoky coal for cooking and heating homes can inhale 10 times higher levels of polycyclic aromatic hydrocarbons (PAH, compounds formed in many burning organic substances, including smoky coal) than someone who smokes 20 cigarettes a day.

Objectives:

* Determine the health effects of smoky coal in Xuan Wei and Fu Yuan counties in China's Yun Nan Province
* Determine how different levels of exposure to smoky coal and other types of fuel affect the amount of smoky coal emissions that are absorbed into the body
* Determine genetic risk factors for lung cancer in the study population and determine how they interact with smoky coal and PAH exposure.

Eligibility:

* Women from Xuan Wei and Fu Yuan counties between 18 and 79 years of age who have lung cancer and do or do not use smoky coal
* Women from Xuan Wei and Fu Yuan counties between 18 and 79 years of age who do not have lung cancer and do or do not use smoky coal

Design:

-Exposure assessment study for users of smoky coal - 150 households

Use of air badges, monitors, and dermal badges to determine subjects' exposure to smoky coal

Collection of blood, urine, cheek cell and sputum samples to measure the amount of smoky coal emissions absorbed into the body and evaluate the types of biologic changes they cause

Interview subjects about their health and family history, occupational exposures, lifestyle factors (e.g., tobacco smoking and diet), and inherited differences in genes

-Case-control study - 1,000 women

Collection of blood, urine, cheek cell and sputum samples to measure how amount of smoky coal emissions absorbed into the body and evaluate types of biologic changes they cause

Interview subjects about their health and family history, occupational exposures, lifestyle factors (e.g., tobacco smoking and diet), and inherited differences in genes

Gene analysis to determine if a genetic variation is associated with an increased or decreased risk of health effects from smoky coal exposure

DETAILED DESCRIPTION:
Females in Xuan Wei County are almost all non-smokers, yet they have the highest lung cancer rate in China. Non-smoking women in Xuan Wei who use smoky coal in their home can inhale ten times higher levels of PAHs than a 20 cigarette per day active smoker, and air concentrations approach levels experienced by workers on the top-side of coke ovens. Several lines of research have provided strong support that the excess lung cancer in this region is caused primarily by PAHs derived from smoky coal exposure. As such, this region of China provides one of the best opportunities in the world to carry out a model study of gene-environment interactions in lung cancer. We have designed a hospital-based case-control study of 500 lung cancer cases and 500 controls among non-smoking women, with controls to be selected through a randomized recruitment design to achieve balance for the main effects of smoky coal exposure and ultimately greater power to detect interactions. The study will be carried out over a three-year period in Xuan Wei and Fu Yuan Counties in Yun Nan Province, China. In addition, we will be carrying out an exposure assessment study (n=150 households) to evaluate air and dermal exposure to PAHs from smoky coal use in order to model PAH exposure experienced by subjects in the case-control study. We will collect buccal cell, sputum, blood, and urine samples from all subjects. The primary goal of the study is to characterize genetic risk factors at the DNA level for lung cancer in this population and determine how they interact with smoky coal and PAH exposure. In addition, the hospital-based design will enable us to collect venous blood samples and cryopreserve lymphocytes, which will allow us to carry out state-of-the-art functional susceptibility assays such as testing ability to repair PAH-damaged DNA and apoptotic capacity, and to measure integrative markers of genomic stability such as telomere length and oxidative damage in mitochondrial DNA. These types of assays have never been conducted in this population and hold great promise to provide insights into cancer risk that will compliment those obtained by genotyping. This study will provide an important complement to and contrast with both DCEG and extramural studies of tobacco smoking and lung cancer, where unraveling the genetic component is challenging in part because hundreds of tobacco carcinogens in various combinations likely contribute.

ELIGIBILITY:
* Cases: Life-long female residents of Xuan Wei and Fu Yuan Counties aged 18 to 79 years are considered the base population. Newly diagnosed primary female lung cancer cases (ICD-9 162), each diagnosis based on a minimum of clinical symptoms, chest X-ray, and a CT scan, will be identified at two hospitals in Xuan Wei County, one hospital in Fu Yuan County, and two hospitals in Qujing District.

Controls: Females alive during the study period who do not have lung cancer and who are residents of Xuan Wei or Fu Yuan Counties aged 18 to 79 will be eligible for recruitment into the study. Diagnosed conditions known to be unrelated to smoky coal exposure or air pollution will be eligible for inclusion into the study. Potential controls diagnosed during the current admission with any cancer or any of the following non-cancer conditions - (respiratory tuberculosis (ICD-10: A15, 16, 19, B90), respiratory infection (A31), neoplasm (C00-D48), ischaemic heart disease (I20-I25), arterial disease (I70-I73), respiratory disease (J00-J99), peptic ulcer (K25-K27), and respiratory symptoms (R04, R06, R09), will be excluded.

Ages: 18 Years to 79 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population is the non-smoking women lived in Xuanwei and Fuyuan, Yunnan Province of China, a region with high lung cancer incidence.
Sampling Method: Probability Sample
Enrollment: 3720 (Actual)
Dates: Start 2006-02-06 (Actual); Primary Completion 2020-11-20 (Actual); Study Completion 2020-11-20 (Actual)

PRIMARY OUTCOMES:
Response-gradient for PAH exposure and lung cancer risk | 2006-2034
  Outcome from this study will include the observation of response-gradient for PAHs exposure due to indoor burning biomass and risk of lung cancer.
Genetic polymorphisms in genes related to PAH metabolism, cell cycle control, and DNA repair associated with the risk of lung cancer | 2006-2034
  Outcome will involve discovering genes related to lung cancer risks among non-smoking Asian women.
Whether polymorphisms in genes related to PAH metabolism, cell cycle control, and DNA repair modify the PAHs-lung cancer association | 2006-2034
  Outcome will also involve the GXE analysis to explore the interaction between genetic factors and environmental exposure.

CONTACTS AND LOCATIONS:
Overall Officials: Qing Lan, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (4):
- China (4):
  - The University of Hong Kong, Hong Kong
  - Kunming Medical University, Kunming
  - China Medical University, Shenyang
  - National University of Singapore, Singapore